CLINICAL TRIAL: NCT00028756
Title: Randomized Phase III Trial Comparing Immediate Versus Deferred Chemotherapy After Radical Cystectomy in Patients With pT3-pT4, and/or N+M0 Transitional Cell Carcinoma (TCC) of the Bladder
Brief Title: Comparison of Immediate and Delayed Adjuvant Chemotherapy in Treating Patients Who Have Undergone a Radical Cystectomy for Stage III or Stage IV Transitional Cell Carcinoma of the Bladder Urothelium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Groupe D'Etude des Tumeurs Uro-Genitales (Other); Institute of Cancer Research, United Kingdom (Other); NCIC Clinical Trials Group (Network); Arbeitsgemeinschaft Urologische Onkologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 30994; EORTC-30994; CDR0000069130; CAN-NCIC-EORTC-30994; ACOSOG-EORTC-30994; NCRI-BLADDER-EORTC-30994; UKCCCR-EORTC-30994; FNCLCC-GETUG-EORTC-30994; N02CM62212 (NIH); 2005-003741-13 (EudraCT Number)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Doxorubicin; Gemcitabine; Vinblastine; Methotrexate; merphos; Cisplatin; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (2):
- Arm I (immediate chemotherapy) (Active Comparator): Beginning within 90 days of radical cystectomy, patients receive a total of 4 courses of adjuvant chemotherapy.
  Interventions: Drug: doxorubicin hydrochloride; Drug: gemcitabine hydrochloride; Drug: vinblastine sulfate; Drug: methotrexate; Drug: cisplatin; Biological: filgrastim
- Arm II (deferred chemotherapy) (Experimental): Beginning at the time of clinical relapse, patients receive a total of 6 courses of adjuvant chemotherapy.
  Interventions: Drug: doxorubicin hydrochloride; Drug: gemcitabine hydrochloride; Drug: vinblastine sulfate; Drug: methotrexate; Drug: cisplatin; Biological: filgrastim

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: vinblastine sulfate — Given IV
  Other Names: 29060-LE; Exal; Velban; Velbe; Velsar
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
Randomized phase III trial to compare the effectiveness of immediate adjuvant chemotherapy with that of adjuvant chemotherapy given when the cancer returns in treating patients who have undergone a radical cystectomy for stage III or stage IV transitional cell carcinoma of the bladder urothelium. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them after surgery may kill any remaining tumor cells. It is not yet known if adjuvant chemotherapy is more effective when given immediately after radical cystectomy (surgery to remove the bladder) or when the cancer returns.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the overall and progression-free survival of patients with stage III or IV transitional cell carcinoma of the bladder urothelium treated with immediate versus deferred adjuvant chemotherapy after radical cystectomy.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, tumor status (pT1-2 vs pT3 vs pT4), and node status (node positive vs node negative with 15 or more nodes sampled vs node negative with less than 15 nodes sampled). Patients are randomized to one of two treatment arms.

ARM I: Beginning within 90 days of radical cystectomy, patients receive a total of 4 courses of adjuvant chemotherapy.

ARM II: Beginning at the time of clinical relapse, patients receive a total of 6 courses of adjuvant chemotherapy.

Patients in both arms receive one of the following chemotherapy regimens to be determined by participating center:

REGIMEN A (Classical M-VAC): Patients receive classical M-VAC comprising methotrexate IV on days 1, 15 and 22; vinblastine IV on days 2, 15, and 22; and doxorubicin IV and cisplatin IV on day 2. Courses repeat every 28 days.

REGIMEN B (High-dose M-VAC): Patients receive high-dose M-VAC comprising methotrexate IV on day 1 and vinblastine IV, doxorubicin IV, and cisplatin IV on day 2. Patients also receive filgrastim (G-CSF subcutaneously once daily on days 4-10. Courses repeat every 14 days.

REGIMEN C (Gemcitabine and cisplatin): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 followed by cisplatin IV on day 1 or 2. Courses repeat every 28 days.

Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK and EORTC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell carcinoma of the bladder urothelium

  * T3-4, N1-3, M0
* No pure squamous cell or adenocarcinoma tumors
* No more than 90 days since prior radical cystectomy and bilateral lymphadenectomy without evidence of microscopic residual disease
* Performance status - WHO 0-1
* WBC at least 3,500/mm^3
* Platelet count at least 120,000/mm^3
* SGOT/SGPT less than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN
* Bilirubin normal
* Glomerular filtration rate greater than 60 mL/min
* No clinically significant cardiac arrhythmia
* No congestive heart failure
* No complete bundle branch block
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study
* Considered fit for cisplatin-containing combination chemotherapy
* No clinically abnormal auditory function
* No known hypersensitivity to E. coli-derived drug preparations
* No grade 2 or greater peripheral neuropathy
* No other prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix, treated basal cell skin cancer, or treated incidental prostate cancer (pT2, Gleason score no greater than 6, and PSA less than 0.5 ng/mL)
* No psychological, familial, sociological, or geographical condition that would preclude study involvement
* No prior systemic chemotherapy
* No prior radiotherapy to the bladder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2001-10; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Duration of survival | 5 years
  Estimated using the Kaplan-Meier technique and compared based on a two sided logrank test with retrospective stratification for the participating cooperative group, the chemotherapy regimen, the T category and the nodal status.
Duration of progression-free survival | 5 years
  Estimated using the Kaplan-Meier technique and compared based on a two sided logrank test with retrospective stratification for the participating cooperative group, the chemotherapy regimen, the T category and the nodal status.

CONTACTS AND LOCATIONS:
Overall Officials: Cora Sternberg, Dr., Study Chair — San Camillo Forlanini Hospitals

REFERENCES:
- [Derived] Sternberg CN, Skoneczna I, Kerst JM, Albers P, Fossa SD, Agerbaek M, Dumez H, de Santis M, Theodore C, Leahy MG, Chester JD, Verbaeys A, Daugaard G, Wood L, Witjes JA, de Wit R, Geoffrois L, Sengelov L, Thalmann G, Charpentier D, Rolland F, Mignot L, Sundar S, Symonds P, Graham J, Joly F, Marreaud S, Collette L, Sylvester R; European Organisation for Research and Treatment of Cancer Genito-Urinary Cancers Group; Groupe d'Etude des Tumeurs Urogenitales; National Cancer Research Institute Bladder Cancer Study Group; National Cancer Institute of Canada Clinical Trials Group; German Association of Urologic Oncology. Immediate versus deferred chemotherapy after radical cystectomy in patients with pT3-pT4 or N+ M0 urothelial carcinoma of the bladder (EORTC 30994): an intergroup, open-label, randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):76-86. doi: 10.1016/S1470-2045(14)71160-X. Epub 2014 Dec 11. PMID 25498218
- See also: Related Info — http://www.eortc.be/clinicaltrials/details.asp?protocol=30994